CLINICAL TRIAL: NCT03780829
Title: Repetitive Acute Intermittent Hypoxia for Spinal Cord Repair
Brief Title: AIH for Spinal Cord Repair
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2848-R
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: SCI
Keywords: spinal cord injury; hypoxia; plasticity
MeSH Terms: conditions — Spinal Cord Injuries; Hypoxia | interventions — Cycloserine; Exercise

STUDY DESIGN:
Intervention Model Description: repetitive intermittent hypoxia treatment combined with exercise and/or NMDA agonist
Who Masked: Participant, Investigator
Masking Description: participants and some research personnel will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- hypoxia plus training (Experimental): combined hypoxia treatment with exercise training
  Interventions: Behavioral: hypoxia; Behavioral: exercise training
- sham hypoxia plus training (Sham Comparator): combined sham hypoxia treatment with exercise training
  Interventions: Behavioral: sham hypoxia; Behavioral: exercise training
- hypoxia plus training plus NMDA agonist (Experimental): combined hypoxia treatment with exercise training and with NMDA agonist treatment
  Interventions: Behavioral: hypoxia; Drug: D-cycloserine; Behavioral: exercise training
- hypoxia plus training plus sham NMDA agonist (Placebo Comparator): combined hypoxia treatment with exercise training and with sham NMDA agonist treatment
  Interventions: Behavioral: hypoxia; Drug: sham-NMDA agonist; Behavioral: exercise training

INTERVENTIONS:
Behavioral: hypoxia — intermittent cycles of normoxia-hypoxia
  Arms: hypoxia plus training; hypoxia plus training plus NMDA agonist; hypoxia plus training plus sham NMDA agonist
Behavioral: sham hypoxia — intermittent cycles of sham hypoxia
  Arms: sham hypoxia plus training
Drug: D-cycloserine — NMDA agonist treatment
  Other Names: NMDA agonist
  Arms: hypoxia plus training plus NMDA agonist
Drug: sham-NMDA agonist — sham-NMDA agonist treatment
  Arms: hypoxia plus training plus sham NMDA agonist
Behavioral: exercise training — bimanual massed practice training

SUMMARY:
Contusive cervical spinal cord injury (cSCI) impairs upper limb function (reach-and-grasp) which limits daily-life activities and thus decreases the quality of life. Promoting neuroplasticity may support upper limb recovery after SCI. Repetitive exposure to acute intermittent hypoxia (rAIH) combined with motor training promotes recovery of motor function after SCI; however, the overall effects of rAIH/training are limited. The investigators will use an adult rat model of long-term contusive cSCI to study novel approaches to enhance the effect of rAIH/training on forelimb function and study the neuronal substrate underlying the effects. The findings will be used to direct the development of more effective rAIH/training approaches for people with contusive, functionally incomplete, cSCI. Because deficits in upper limb function are a major problem after stroke, amyotrophic lateral sclerosis, multiple sclerosis, and other motor disorders, this work may also be relevant for patients with other types of central nervous system (CNS) lesions.

DETAILED DESCRIPTION:
The overall goal is to develop effective, clinically applicable, approaches to restore upper limb function (reach-and-grasp) after chronic contusive cervical spinal cord injury (cSCI). Impairments in upper limb function significantly reduce the quality of life for people with cSCI. Reach-and-grasp actions in animals and humans are largely controlled by the corticospinal tract (CST). The investigators argue that promoting plasticity within the CST may support the recovery of upper limb function after cSCI. Repetitive exposure to acute intermittent hypoxia (rAIH) combined with motor training is a safe, minimally invasive, treatment that elicits neuroplasticity resulting in improved recovery after cSCI, but its overall effects remain limited. The main goals are to: 1) enhance rAIH/training-induced aftereffects on forelimb function and increase the understanding of the neuronal substrates in an adult rat model of chronic contusive cSCI, and 2) use this knowledge to guide the development of more effective rAIH/training approaches to improve upper limb function in humans with chronic contusive cSCI.

In Specific Aim 1, using an adult rat model of chronic contusive cSCI, the investigators will investigate the effects of rAIH frequency and dose on rAIH/training-mediated functional recovery of the impaired forelimb. Also, the investigators will combine rAIH/training with N-methyl-D-aspartate receptor (NMDA)-mediated synaptic plasticity through D-cycloserine treatment and study the effects on recovery of forelimb function. Immunocytochemistry with imaging techniques will be used to assess structural neuronal plasticity in the CST after rAIH/training. In Specific Aim 2, in people with chronic incomplete cSCI, guided by the findings in Specific Aim 1, the investigators will study the effects of rAIH frequency and concurrent D-cycloserine treatment on rAIH/training-mediated upper limb function recovery. The investigators will comprehensively analyze the effects of rAIH on the strength of electrophysiological and functional aftereffects in the upper limb.

The proposed research will provide new knowledge on rAIH/training-mediated functional and anatomical aftereffects (Specific Aim 1), which will be used to develop effective rAIH/training protocols for people with contusive, functionally incomplete, cSCI (Specific Aim 2). The data from the investigators' experiments may lead to clinically applicable approaches that improve arm and hand function recovery after chronic contusive cSCI, which would positively impact the quality of life of Veterans with cSCI. The relevance of this proposal is emphasized by the limited efficacy of current strategies to improve upper limb function after cSCI.

ELIGIBILITY:
Inclusion Criteria:

* Male and females Veterans between 18-85 years
* Chronic cSCI (1 yr of injury)
* Cervical injury at C8 or above
* Sensory function: impaired (score of 1) but not absent (score of 0) or intact (score of 2) innervations in dermatomes C6, C7 and C8 during light touch and pin prick stimulus using the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) sensory scores
* Motor function: Able to grasp small objects with one hand and able to perform a visible precision grasp between the index finger and thumb
* Motor scores ISNCSCI: 1 to 4 but not 5 on finger flexors and finger abductors on the hand tested.

  * These criteria were selected to ensure that hand impairment will not interfere with the ability to perform training and proposed tests

Inclusion criteria for controls:

* Male and females (18-80 years)
* Right handed
* Able to complete precision and power grips

Exclusion Criteria:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs

  * chlorpromazine
  * clozapine
  * or tricyclic antidepressants
* Pregnant females
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease as spinal stenosis, spina bifida or herniated cervical disk
* AIH Exclusion Criteria (in addition to the above listed exclusion criteria):

  * resting heart rate > 120 bpm
  * resting systolic blood pressure >180 mmHg
  * resting diastolic blood pressure >100 mmHg
  * self-reported history of unstable angina or myocardial infarction within the previous month
  * resting SpO2 > or equal to 95%
  * cardiopulmonary complications such as COPD

Exclusion criteria for healthy controls:

* Same as for SCI individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Change in grip strength | baseline, 1st week, 2nd week, 4th week, 8th week, and 12th week
  Grip strength will be measured using a hand-held dynamometer, with an average force (measured in dynes) taken over the course of three trials. A rest break is provided between trials. Strength testing will be completed bilaterally.
Change in pinch strength | baseline, 1st week, 2nd week, 4th week, 8th week, and 12th week
  Pinch strength will be assessed using a digital pinch gauge (unit of Force= Newton). The minimum value of zero will be assigned when a participant cannot actively squeeze the pinch meter between the thumb and index finger. The mean value of total of 3 trials will be assessed, with a rest break provided between trials.
Change in motor evoked potential size | 30 minutes before and 30 minutes after intervention
  Resting and active motor thresholds (RMT and AMT) will be tested in each of the muscles using a stimulator.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Oudega, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No